CLINICAL TRIAL: NCT04331652
Title: Bipolar 15 Charrières (Ch.) Office Resectoscope : Polypectomy Without Anesthesia - Prospective Evaluation
Brief Title: Bipolar 15 Charrières Office Resectoscope : Polypectomy Without Anesthesia
Acronym: HSC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: change of practices
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019_0026
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Polyps Uterus
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Polypectomy without anesthesia or analgo-sedation (Experimental): Patient will undergo polypectomy without anesthesia.
  Interventions: Procedure: Polypectomy without anesthesia or analgo-sedation

INTERVENTIONS:
Procedure: Polypectomy without anesthesia or analgo-sedation — Premedication: paracetamol 1g oral. Patient will undergo polypectomy without anesthesia. During the procedure, pain will be monitored using a pain assessment scale from 0 to 10 (0 meaning no pain and 10 meaning maximum pain imaginable). At any time, if the patient express a pain strictly superior to 4 an analgo-sedation will be proposed and/or general anesthesia.
  Pulse and blood pressure will be monitored. Assessment of patient satisfaction after the intervention.

SUMMARY:
This study aimed to the feasibility of polypectomy without anesthesia using a 15 Ch. resectoscope in women with uterine polyps.

DETAILED DESCRIPTION:
Endometrial polyps are frequent gynecological pathologies leading to metrorrhagia, infertility, miscarriages and the risk of transformation into malignant pathology. The discovery of an endometrial polyp requires its removal.

The treatment of endometrial polyps is conventionally carried out by hysteroscopic resection under general anesthesia with a bipolar resector of 22 Charrières (Ch) or more after dilation of the uterine cervix in the operating room.

Following the recent appearance of a 15 Ch. bipolar mini-resectoscope, it seems that uterine dilation and anesthesia could be avoided by reducing the caliber of the instrument.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 or over
* Patients with 1 to 2 endometrial polyps
* Polyps diagnosed by ultrasound and / or diagnostic hysteroscopy following a check-up for menometrorrhagia, infertility or during a check-up
* Polyps measuring less than 3 cm
* Have signed a consent form
* Be affiliated with a Health Insurance plan.

Exclusion Criteria:

* Pregnant or lactating patient
* Cervical stenosis
* Patient having more than 2 polyps
* Polyps measuring 3 cm or more
* Malignant cells on histology
* Associated indication of endometrectomy or other endo-uterine gesture
* Hypersensitivity to remifentanil or to other fentanyl derivatives or to any of the excipients of the specialty used
* Hypersensitivity to propofol or to any of the excipients of the specialty used
* Cardiac pathology
* Diaphragmatic hernia
* Morbid obesity (BMI> 35)
* Invasive cervical cancer
* Chronic obstructive pulmonary disease
* Patient presenting a strictly greater than 4 on a pain scale (from 0 to 10) during a diagnostic hysteroscopy
* Does not speak and / or understand French
* Be deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patient with uterin polyp(s)
Enrollment: 13 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of polypectomy, with a mini-resectoscope of 15 bipolar careers, without general anesthesia or analgo-sedation | 1 day (surgery)
  Use or not of general anesthesia or analgo-sedation during the surgery

SECONDARY OUTCOMES:
Pain assessment during and after surgery | 1 day (surgery)
  Pain assessment on a scale from 0 to 10; before surgery, during surgery (during the introduction of the hysteroscope into the uterine cavity, during the possible placement of a speculum and during the removal of the polyp at the handle) then 15 minutes, 1 hour and 2 hours post-operative
Capacity and clinical condition of the patient allowing her discharge | 1 day (surgery)
  Capacity and clinical condition of the patient allowing her discharge 15 minutes, 1 hour and 2 hours after surgery
Patient satisfaction | 4 months
  Patient satisfaction on a scale from 1 to 5 (1 meaning not satisfied at all and 5 very satisfied)
Post operative diagnostic hysteroscopy result | 4 months
  Control diagnostic hysteroscopy: success if absence of visible intra-cavitary projection at the base of the excised polyp(s)
Identification of factors influencing the success of the main criterion | 4 months
  Correlations between preoperative data and main evaluation criterion (patient with or without analgo-sedation and or general anesthesia)

CONTACTS AND LOCATIONS:
Overall Officials: Angeline FAVRE-INHOFER, Dr, Principal Investigator — Hopital Foch; Marie Carbonnel, Dr, Study Director — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No